CLINICAL TRIAL: NCT01672047
Title: Effect of Vitamin D Supplementation on Coronary Calcification and Parathyroid Hormone in CKD Patients
Acronym: EVIDENCE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Wang Mei, Professor, Peking University People's Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PURCP201103
Record Dates: First submitted 2012-08-21; First posted 2012-08-24 (Estimated); Last update posted 2012-08-30 (Estimated); Status verified 2012-08

CONDITIONS: Chronic Kidney Disease; Vitamin D Deficiency
Keywords: The 25(OH) vitamin D level; The 1.25(OH) vitamin D level; The intact PTH level; The calcification score of coronary artery; The microalbuminuria level
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Ergocalciferols

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treament (Experimental): Intervention Vitamin D2
  Interventions: Drug: Vitamin D2
- Control (No Intervention): Not take Vitamin D2

INTERVENTIONS:
Drug: Vitamin D2 — 25（OH）D level <12 nmol/L 50000IU/weekX12week， 12-39 nmol/L 50000IU/weekX4week then，50000IU/month， 40-75 nmol/L 50000IU/month， 75-116.75nmol/L 25000IU/month， >116.75nmol/L stopped.
  Other Names: Vitmain D2 capsule
  Arms: Treament

SUMMARY:
The investigators hypothesize that the chronic kidney disease patients who suffer from vitamin D deficiency will be benefit from given Vitamin D2 because coronary artery calcification and hyperparathyroidism will be improved.

DETAILED DESCRIPTION:
We will call for 350 CKD patients (250 CKD3-5stage and 100 CKD5D stage)who suffer from vitamin D deficiency.They will be divided into 2 groups. One group will be given vitamin D and the other will not. They will take coronary artery CT test every year(in 2 years).We will compare the coronary calcification progression between the 2 groups.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease patients (3-5D)
* serum 25（OH）D < 40nmol/L(16ng/ml)，serum calcium < 2.55mmol/L（10.2mg/dL）；
* willing to sign
* could obey the follow up design

Exclusion Criteria:

* allergy to vitamin D
* heart failure (NYHA more than 2 grade)
* pregnant
* malignant tumor
* critical hepatic disease
* taking Vitamin D or analogue in 3 recent months
* taking other clinical trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2012-04; Primary Completion 2014-04 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
the improvement of coronary artery calcification | 2 years
  We use CT to detect the coronary artery calcification score in the chronic kidney disease patients for 3 times (baseline, 12 month and 24 month). We will compare the 2 arms （treatment or not）to know if there is any difference。

SECONDARY OUTCOMES:
the improvement of proteinuria | 2 years
  We detect the microalbuminuria in the chronic kidney disease patients for 5 times (baseline, 6 month,12 month 18month and 24 month). We will compare the 2 arms （treatment or not）to know if there is any difference。

CONTACTS AND LOCATIONS:
Overall Officials: Mei Wang, MD, PhD, Principal Investigator — Peking University People's Hospital
Locations (1):
- The People's Hospital of Peking University, Beijing, Beijing Municipality, China